CLINICAL TRIAL: NCT01055613
Title: Investigational Multi-purpose Contact Lens Care Solution.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR-1624
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-07

CONDITIONS: Contact Lens Wear

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental multi-purpose solution (Experimental): Multi-purpose contact lens care solution.
  Interventions: Device: Vistakon Investigational Multi-Purpose Solution I
- ReNu MultiPlus Multi-Purpose Solution (Active Comparator): Multi-purpose contact lens care solution.
  Interventions: Device: ReNu MultiPlus Multi-Purpose Solution

INTERVENTIONS:
Device: Vistakon Investigational Multi-Purpose Solution I — Multi-purpose contact lens care solution.
  Arms: Experimental multi-purpose solution
Device: ReNu MultiPlus Multi-Purpose Solution — Multi-purpose contact lens care solution
  Arms: ReNu MultiPlus Multi-Purpose Solution

SUMMARY:
This study compares an investigational contact lens care multi-purpose solution to a currently marketed multi-purpose solution.

ELIGIBILITY:
Inclusion Criteria:

* must be an adapted contact lens wearer
* best corrected distance visual acuity must be 20/25 or better in each eye
* must be wearing their habitual lenses on a daily wear basis
* must be willing to refrain from swimming during the study

Exclusion Criteria:

* any systemic diseases that may interfere with contact lens wear
* any clinically significant ocular disease
* any ocular infection
* use of certain medications
* any grade 2 or greater slit lamp findings
* any know sensitivity to marketed contact lens care solutions
* currently pregnant or lactating
* monovision corrected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Fresno, California
  - Pismo Beach, California
  - Louisville, Colorado
  - Bloomfield, Connecticut
  - Jacksonville, Florida
  - Overland Park, Kansas
  - East Lansing, Michigan
  - Warrensburg, Missouri
  - Grove City, Ohio
  - Grants Pass, Oregon
  - Kingston, Pennsylvania
  - Sioux Falls, South Dakota
  - Memphis, Tennessee
  - Salt Lake City, Utah
  - Laramie, Wyoming

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 312 subjects were enrolled in this study. Of the enrolled subjects 12 did not meet the eligibility criteria and 300 were randomized to treatment using an allocation of 2:1 for test and control, respectively. Of the 300 randomized subjects 13 were discontinued from the study and 287 subjects completed the study.
Groups:
- Experimental Multi-purpose Solution: Experimental multi-purpose contact lens care solution (Test treatment)
- ReNu MultiPlus Multi-Purpose Solution: Marketed multi-purpose contact lens care solution (Control Treatment).
Period: Overall Study
Arm/Group | Experimental Multi-purpose Solution | ReNu MultiPlus Multi-Purpose Solution
Started | 200 | 100
Completed | 191 | 96
Not Completed | 9 | 4
Not completed — No Longer Meets Eligibility Criteria | 3 | 0
Not completed — Unacceptable lens fit | 1 | 0
Not completed — Discomfort | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Subject Disinterest | 1 | 1

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed a study lens.
Groups:
- Experimental Mutli-purpose Solution: Experimental multi-purpose solution (Test treatment) .
- ReNu Multi-purpose Solution: Marketed multi-purpose solution (Control Treatment).
- Total: Total of all reporting groups
Arm/Group | Experimental Mutli-purpose Solution | ReNu Multi-purpose Solution | Total
Number analyzed (Participants) | 200 | 100 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.40 (9.231) | 31.05 (8.624) | 31.73 (8.928)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 71 | 216
  Male | 55 | 29 | 84
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 5 | 6 | 11
  Native Hawaiian or other Island Pacificer | 0 | 1 | 1
  Asian | 3 | 2 | 5
  White | 185 | 88 | 273
  Other | 6 | 3 | 9
  American Indian or Native Alaskian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 200 | 100 | 300

OUTCOME MEASURES:

1. Primary Outcome: Slit Lamp Findings
Description: Each subjects' eye was examined using a bio-microscope. Slit lamp findings were graded with a 5-point scale (i.e. Grade 0= None, Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). The number of eyes with Grade 3 or higher for each lens was reported for each assessment.
Time Frame: 3 months
Population: The analysis population consists of all subjects that were dispensed a solution during the course of the study.
Measure: Number; unit: Subjects Eyes
Units Other Than Participants: Subject Eye's
Arm/Group | Experimental Multi-purpose Solution | ReNu MultiPlus Multi-Purpose Solution
Number analyzed (Participants) | 191 | 96
Number analyzed (Subject Eye's) | 382 | 192
Subjects Eyes
  Corneal Staining | 11 | 16
  Conjunctival Staining | 0 | 0
  Tarsal Abnormalities | 14 | 12

2. Primary Outcome: Distance Visual Acuity (LogMAR)
Description: Distance visual acuity was collected at the 1-, 2-, 3-week and 1- and 3- month follow-up evaluations. The average LogMAR across all visits for each lens type was reported.
Time Frame: Up to 3 Months
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Subject Eyes
Arm/Group | Experimental Multi-purpose Solution | ReNu MultiPlus Multi-Purpose Solution
Number analyzed (Participants) | 191 | 96
Number analyzed (Subject Eyes) | 382 | 192
LogMAR | -0.030 (0.0639) | -0.031 (0.0634)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 3 months.
Arm/Group | Experimental Multi-purpose Solution | ReNu MultiPlus Multi-Purpose Solution
Serious Adverse Events (participants affected / at risk) | 1/200 | 0/100
Other Adverse Events (participants affected / at risk) | 0/200 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Multi-purpose Solution (N=200) | ReNu MultiPlus Multi-Purpose Solution (N=100)
Microbial Keratitis (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days